CLINICAL TRIAL: NCT04146376
Title: Von Willebrand Factor in Pregnancy (VIP) Study: A Multicenter Study of Wilate Use in Von Willebrand Disease for Childbirth
Brief Title: Von Willebrand Factor in Pregnancy (VIP) Study
Acronym: VIP
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Ergomed (Industry); Octapharma (Industry)
Responsible Party: Principal Investigator, Jill Johnsen, Professor, School of Medicine: Hematology and Oncology, University of Washington
Other Study IDs: STUDY00016309
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Von Willebrand Diseases
Keywords: von Willebrand Disease; von Willebrand Factor; postpartum hemorrhage
MeSH Terms: conditions — von Willebrand Diseases; Postpartum Hemorrhage | interventions — von Willebrand Factor; Tranexamic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma collection for coagulation parameters Whole blood collection for DNA and RNA analysis Cord blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-Corrector: Patients with gestational week 34-38 von Willebrand factor activity, or von Willebrand factor ristocetin cofactor, or Factor VIII procoagulant activity less than 100 percent will be termed non-correctors. When laboratory monitoring can be performed, patients with an isolated von Willebrand factor collagen binding type 2 defect, von Willebrand factor collagen binding less than 100 percent can also be enrolled and determined as a non-corrector.
  Interventions: Other: Use of a postpartum diary and additional blood draws; Drug: VWF replacement therapy with Wilate; Drug: Tranexamic acid
- Corrector: Patients with von Willebrand factor parameter levels greater than or equal to 100 percent self-corrected at gestational weeks 34-38 will be termed correctors.
  Interventions: Drug: Tranexamic acid; Other: Use of a postpartum diary and additional blood draws.

INTERVENTIONS:
Other: Use of a postpartum diary and additional blood draws — A diary will be used to capture postpartum hemorrhage (PPH), Wilate and tranexamic acid use, other drug use, bleeding episodes, and treatment schedules.
  Several blood draws additional to what is expected for routine clinical care will also be taken.
  Groups: Non-Corrector
Drug: VWF replacement therapy with Wilate — This study design uses on-label Wilate for VWF replacement therapy for delivery and the postpartum period in VWD patients whose VWF levels are <100% in the third trimester of pregnancy
  Groups: Non-Corrector
Drug: Tranexamic acid — This study design uses tranexamic acid for prophylaxis for postpartum hemorrhage for all women with VWD
Other: Use of a postpartum diary and additional blood draws. — A diary will be used to capture postpartum hemorrhage (PPH), tranexamic acid use, other drug use, bleeding episodes, and treatment schedules.
  Several blood draws additional to what is expected for routine clinical care will also be taken.
  Groups: Corrector

SUMMARY:
In pregnant women with von Willebrand disease (VWD) who by the third trimester do not have von Willebrand factor (VWF) or factor VIII (FVIII) levels greater than 50-100%, specific guidance is lacking for delivery planning in terms of how high of a VWF level should be achieved to reduce bleeding.

This is a prospective, open-label, cohort study in women with VWD using Wilate VWF replacement therapy to maintain trough or minimum VWF levels of 100-150% for delivery and the immediate postpartum period, followed by levels of 50-100% for 5-10 days after delivery, depending upon the route of delivery. The primary objective is to document the rate of primary postpartum hemorrhage (PPH). The secondary objective is to document further effectiveness outcomes and safety.

DETAILED DESCRIPTION:
For pregnant women with von Willebrand disease (VWD) who by the third trimester do not have von Willebrand factor (VWF) or factor VIII (FVIII) levels > 50-100%, specific guidance is lacking for delivery planning for how high a VWF level should be achieved. Specifically, guidance is lacking on whether VWF replacement therapy should target a VWF minimum level in the 100-150% range, i.e., a range closer to the 200-250% levels observed in normal pregnancy.

This is a prospective, open-label, cohort study using Wilate VWF replacement therapy, trough or minimum VWF levels of 100-150% will be maintained for delivery in women with VWD whose third trimester VWF levels are <100%. This group is termed "non-correctors". Women with VWD whose third trimester VWF levels spontaneously rise to >100% will be assigned to the "corrector" group, and these women will not receive VWF replacement therapy. All patients will receive tranexamic acid for 14 days postpartum. Outcome parameters will be assessed for all patients.

The investigators or qualified research personnel will approach all consecutive pregnant VWD patients until 65 non-corrector patients have completed the study protocol, and up to 30 corrector patients have completed the study protocol. Patients with gestational week 34-38 von Willebrand factor activity (VWF:Act) or von Willebrand factor ristocetin cofactor (VWF:RCo), and/or Factor VIII procoagulant activity (FVIII:C) less than 100 percent will be used to assign patients to the non-corrector group. When VWF collagen binding (VWF:CB) laboratory monitoring can be performed, patients with an isolated VWF:CB type 2 defect can also be enrolled.

Rate of primary postpartum hemorrhage, severe postpartum hemorrhage, secondary postpartum hemorrhage will be measured. Safety and secondary laboratory measures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* von Willebrand Disease (VWD) patients defined prepartum as Type 1 per National Heart, Lung, and Blood Institute (NHLBI) criterion of von Willebrand Factor (VWF) level less than 30 percent, or Type 2, or Type 3 VWD

or

* A diagnosis of VWD and VWF and Factor VIII (FVIII) levels obtained in gestational weeks 34-38 that determine enrollment in the non-corrector group:
* Patients with gestational week 34-38 VWF:Ag, VWF:Act (or VWF:RCo), or FVIII:C less than 100 percent will be enrolled in the non-corrector group. In patients with an isolated VWF:CB type 2 defect, VWF:CB less than 100 percent can also be determined as a non-corrector
* Patients with all VWF parameter levels greater than or equal to 100 percent self-corrected at gestational weeks 34-38 will be enrolled in the corrector group

Written informed consent from the patient prepartum, before gestational week 39

Exclusion Criteria:

* Presence of a clinical contraindication to receive wilate or tranexamic acid, as determined by the health care provider, such as a prior drug reaction
* Presence of other concurrent disorder of hemostasis, platelet dysfunction, or collagen disorders
* Presence of liver disease or renal disease, clinical suspicion or diagnosis of preeclampsia or eclampsia, HELLP syndrome, TTP, DIC, or other acquired vasculopathy or coagulopathy
* Age less than 18 years
* Inability of the local laboratory to monitor the VWF laboratory tests needed during the course of treatment to determine Wilate dosing adjustments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators or qualified research personnel will approach all consecutive pregnant VWD patients. Patients who meet all of the inclusion criteria and none of the exclusion criteria are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2019-10-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
rate of primary postpartum hemorrhage (PPH) | within 24 hours postpartum
  defined as the estimated and/or quantified blood loss greater than or equal to 1000 mL within 24 hours postpartum; unplanned transfusion of blood products related to blood loss in the first 24 hours postpartum.
  As a subset of primary PPH, severe primary PPH is defined as the estimated and/or quantified blood loss greater than or equal to 1500 mL and/or requirement of greater than 2 units packed red blood cells within 24 hours postpartum; primary PPH greater than 1000 mL and evidence of maternal hemodynamic instability (tachycardia, hypotension) and/or end organ damage with no other etiology (oliguria, creatinine greater than 0.8, etc.)

SECONDARY OUTCOMES:
rate of secondary postpartum hemorrhage (PPH) | 24 hours to 6 weeks postpartum
  excessive blood loss: any transfusions not anticipated in the antepartum birth plan and unrelated to a primary PPH, including number and type of blood component units (blood products, red blood cells, plasma, platelets, cryoprecipitate) transfused within 48 hours after diagnosis and management; any transfusions not anticipated in the antepartum birth plan and unrelated to a primary PPH, including number and type of blood component units (blood products, red blood cells, plasma, platelets, cryoprecipitate) transfused beyond 48 hours after diagnosis and management; change in antepartum hemoglobin; change in pictorial blood assessment chart (PBAC) score; number of patients needing pharmacologic or surgical interventions for bleeding (e.g., use of Bakri balloon, angiographic embolization, B-Lynch sutures, surgical arterial ligation, or hysterectomy for persistent bleeding); iron levels (serum iron, TIBC, and ferritin) 6 weeks postpartum

OTHER OUTCOMES:
occurrence of venous or arterial thrombus | up to 42 days postpartum
  clinically documented venous or arterial thrombus
occurrence of infusion-related reactions | up to 42 days postpartum
  clinically documented infusion-related reactions
laboratory assessment of efficacy and VWF replacement | up to 42 days postpartum
  central laboratory assessment of VWF parameters relative to bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Johnsen, M.D., Principal Investigator — University of Washington; Barbara A Konkle, M.D., Principal Investigator — Washington Center for Bleeding Disorders; Peter A Kouides, M.D., Principal Investigator — Mary M. Gooley Hemophilia Center
Locations (11):
- United States (11):
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Bleeding & Clotting Disorders Institute, Peoria, Illinois
  - Tulane University School of Medicine, Louisiana Center for Bleeding and Clotting Disorders, New Orleans, Louisiana
  - Oregon Health & Science University, Portland, Oregon
  - The Pennsylvania State University, Hershey, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Washington Center for Bleeding Disorders, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James AH, Konkle BA, Kouides P, Ragni MV, Thames B, Gupta S, Sood S, Fletcher SK, Philipp CS. Postpartum von Willebrand factor levels in women with and without von Willebrand disease and implications for prophylaxis. Haemophilia. 2015 Jan;21(1):81-7. doi: 10.1111/hae.12568. Epub 2014 Oct 21. PMID 25333737
- [Background] Drury-Stewart DN, Lannert KW, Chung DW, Teramura GT, Zimring JC, Konkle BA, Gammill HS, Johnsen JM. Complex changes in von Willebrand factor-associated parameters are acquired during uncomplicated pregnancy. PLoS One. 2014 Nov 19;9(11):e112935. doi: 10.1371/journal.pone.0112935. eCollection 2014. PMID 25409031
- [Background] Kouides PA. Present day management of inherited bleeding disorders in pregnancy. Expert Rev Hematol. 2016 Oct;9(10):987-95. doi: 10.1080/17474086.2016.1216312. Epub 2016 Aug 2. PMID 27459638
- [Background] Abbassi-Ghanavati M, Greer LG, Cunningham FG. Pregnancy and laboratory studies: a reference table for clinicians. Obstet Gynecol. 2009 Dec;114(6):1326-1331. doi: 10.1097/AOG.0b013e3181c2bde8. PMID 19935037
- [Background] Szecsi PB, Jorgensen M, Klajnbard A, Andersen MR, Colov NP, Stender S. Haemostatic reference intervals in pregnancy. Thromb Haemost. 2010 Apr;103(4):718-27. doi: 10.1160/TH09-10-0704. Epub 2010 Feb 19. PMID 20174768
- [Background] Huq FY, Kulkarni A, Agbim EC, Riddell A, Tuddenham E, Kadir RA. Changes in the levels of factor VIII and von Willebrand factor in the puerperium. Haemophilia. 2012 Mar;18(2):241-5. doi: 10.1111/j.1365-2516.2011.02625.x. Epub 2011 Sep 28. PMID 21951573
- [Background] Nichols WL, Hultin MB, James AH, Manco-Johnson MJ, Montgomery RR, Ortel TL, Rick ME, Sadler JE, Weinstein M, Yawn BP. von Willebrand disease (VWD): evidence-based diagnosis and management guidelines, the National Heart, Lung, and Blood Institute (NHLBI) Expert Panel report (USA). Haemophilia. 2008 Mar;14(2):171-232. doi: 10.1111/j.1365-2516.2007.01643.x. PMID 18315614
- [Background] Demers C, Derzko C, David M, Douglas J; Society of Obstetricians and Gynecologists of Canada. Gynaecological and obstetric management of women with inherited bleeding disorders. J Obstet Gynaecol Can. 2005 Jul;27(7):707-32. doi: 10.1016/s1701-2163(16)30551-5. English, French. PMID 16100628
- [Background] Mannucci PM, Franchini M, Castaman G, Federici AB; Italian Association of Hemophilia Centers. Evidence-based recommendations on the treatment of von Willebrand disease in Italy. Blood Transfus. 2009 Apr;7(2):117-26. doi: 10.2450/2008.0052-08. PMID 19503633
- [Background] Laffan MA, Lester W, O'Donnell JS, Will A, Tait RC, Goodeve A, Millar CM, Keeling DM. The diagnosis and management of von Willebrand disease: a United Kingdom Haemophilia Centre Doctors Organization guideline approved by the British Committee for Standards in Haematology. Br J Haematol. 2014 Nov;167(4):453-65. doi: 10.1111/bjh.13064. Epub 2014 Aug 12. No abstract available. PMID 25113304
- [Background] Stoof SC, van Steenbergen HW, Zwagemaker A, Sanders YV, Cannegieter SC, Duvekot JJ, Leebeek FW, Peters M, Kruip MJ, Eikenboom J. Primary postpartum haemorrhage in women with von Willebrand disease or carriership of haemophilia despite specialised care: a retrospective survey. Haemophilia. 2015 Jul;21(4):505-12. doi: 10.1111/hae.12635. Epub 2015 Feb 16. PMID 25688733
- [Background] Hawke L, Grabell J, Sim W, Thibeault L, Muir E, Hopman W, Smith G, James P. Obstetric bleeding among women with inherited bleeding disorders: a retrospective study. Haemophilia. 2016 Nov;22(6):906-911. doi: 10.1111/hae.13067. Epub 2016 Oct 5. PMID 27704714
- [Background] Janssen CA, Scholten PC, Heintz AP. A simple visual assessment technique to discriminate between menorrhagia and normal menstrual blood loss. Obstet Gynecol. 1995 Jun;85(6):977-82. doi: 10.1016/0029-7844(95)00062-V. PMID 7770270
- [Background] James AH, Jamison MG. Bleeding events and other complications during pregnancy and childbirth in women with von Willebrand disease. J Thromb Haemost. 2007 Jun;5(6):1165-9. doi: 10.1111/j.1538-7836.2007.02563.x. PMID 17403089
- [Background] Kirtava A, Drews C, Lally C, Dilley A, Evatt B. Medical, reproductive and psychosocial experiences of women diagnosed with von Willebrand's disease receiving care in haemophilia treatment centres: a case-control study. Haemophilia. 2003 May;9(3):292-7. doi: 10.1046/j.1365-2516.2003.00756.x. PMID 12694520
- [Background] Govorov I, Lofgren S, Chaireti R, Holmstrom M, Bremme K, Mints M. Postpartum Hemorrhage in Women with Von Willebrand Disease - A Retrospective Observational Study. PLoS One. 2016 Oct 25;11(10):e0164683. doi: 10.1371/journal.pone.0164683. eCollection 2016. PMID 27780267
- [Background] James AH, Cooper DL, Paidas MJ. A global quantitative survey of hemostatic assessment in postpartum hemorrhage and experience with associated bleeding disorders. Int J Womens Health. 2017 Jul 3;9:477-485. doi: 10.2147/IJWH.S132135. eCollection 2017. PMID 28740434
- [Background] Kujovich JL. von Willebrand disease and pregnancy. J Thromb Haemost. 2005 Feb;3(2):246-53. doi: 10.1111/j.1538-7836.2005.01150.x. No abstract available. PMID 15670029